CLINICAL TRIAL: NCT01588249
Title: A Novel Formulation of Pasteurized Maple Cough Syrup Compared With Placebo on Nocturnal Cough and Sleep Quality in Infants With Upper Respiratory Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Revisiting product options
Sponsor: Zarbee's Inc. (Industry)
Collaborators: Advanced Clinical Research Services, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZMCS-6441
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Cough; Upper Respiratory Infection; Nocturnal Cough
MeSH Terms: conditions — Cough; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Novel formulation of pasteurized maple cough syrup (Experimental)
  Interventions: Dietary Supplement: Pasteurized maple syrup
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pasteurized maple syrup
  Arms: Novel formulation of pasteurized maple cough syrup
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Cough is a frequent symptom in children and infants and is one of the most common reasons parents visit a healthcare provider for their child. The US Food and Drug Administration has issued a warning that over-the-counter cough and cold medicines including antihistamines, decongestants, anti-tussives, and expectorants should not be administered to children younger than 2 years of age due not only to lack of proven efficacy, but also because of important safety concerns. A product that has been used in alternative medicine for cough is maple syrup. Although no studies have formally evaluated the use of maple syrup for nocturnal cough associated with URI, the demulcent effect of maple syrup may provide some relief from cough in children. A novel formulation of pasteurized maple cough syrup, when compared to placebo, should provide superior relief on nocturnal cough and the sleep difficulty associated with URI in children under 12 months and sleep difficulty of their parent/caregiver.

ELIGIBILITY:
Inclusion Criteria

1. Otherwise healthy male or female infant who is between 0 and 12 months of age.
2. Presents to clinic with a URI characterized by the presence of rhinorrhea and cough for 7 or fewer days' duration.
3. Patient is an appropriate candidate, in the judgment of the investigator, to participate in the study.
4. Parents/caregivers provide an answer of at least "somewhat" (3 points on a 7-point Likert scale) for a minimum of 2 of the 3 questions related to nocturnal cough frequency, effect on child's sleep, and effect on parental/caregiver sleep based on the previous night's symptoms (see Section 11.0).
5. Parent/legal authorized representative provides written informed consent for child to participate in study.
6. Parent/caregiver who is willing and able to comply with study requirements.

Exclusion Criteria

1. Signs or symptoms of a more treatable disease (eg, asthma, pneumonia, laryngotrachebronchitis, sinusitis, allergic rhinitis).
2. Diagnosis of influenza, bronchiolitis or respiratory syncytial virus (RSV).
3. History of reactive airways disease, asthma, or chronic lung disease.
4. Use of any medication to treat cough within 6 hours of bedtime on the evening prior to or on the day of enrollment. (Use of analgesic medications such as acetaminophen or ibuprofen is not exclusionary.)
5. Presence of any significant disease including immunodeficiency, hepatic, renal, cardiovascular, or hematologic disease or any other health condition that, in the opinion of the investigator, would preclude participation in the study.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cough frequency between the first night and the end of the second night. | baseline and day 2

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Willow Creek Pediatrics, Draper, Utah
  - Families First Pediatrics, South Jordan, Utah
  - Southwest Children's Clinic, West Jordan, Utah